CLINICAL TRIAL: NCT01514799
Title: Randomized Study Comparing the Effects of Gastric Bypass Using a Long BP-limb vs. a Long Alimentary Limb in Morbid Obesity
Brief Title: Effects of Long Biliopancreatic Limb vs. Long Alimentary Limb in Superobesity, a Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aleris Obesity (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011_HG_Aleris_limb_length
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Morbid Obesity; Weight Loss
Keywords: gastric bypass; morbid obesity; gut function; weight loss
MeSH Terms: conditions — Obesity, Morbid; Weight Loss | interventions — Gastric Bypass

STUDY DESIGN:
Intervention Model Description: Randomised study between long and standard biliopancreatic limb in gstric bypass surgery
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomisation in the OR, (closed envelopes, blocks of six) no further info to ward or follow-up unit. No specific info as to randomisation outcome given to patients, all patients follow same protocol.
  Code number in operative charts.
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard length bp limb, long alimentary limb (Active Comparator): our normal way of doing a gastric bypass 60 cm BP limb
  Interventions: Procedure: gastric bypass
- Long BP limb (Experimental): 200 cm BP limb
  Interventions: Procedure: gastric bypass

INTERVENTIONS:
Procedure: gastric bypass — two techniques of gastric bypass for studying the effects of making a long BP-limb

SUMMARY:
Super Obesity, i.e. a BMI above 50, is difficult to treat. Normal gastric bypass surgery is not always enough for proper weight control. Bypassing a longer segment of the gut may be more beneficial. Which part to bypass is not clear.

The investigators want to compare the effects between preventing a 60 cm proximal (oral) portion of the jejunum from food contact with the effects when preventing a 200 cm part of the jejunum from contact with bile and pancreatic juice.

Endpoints are quality of life, gastrointestinal function, and weight development.

DETAILED DESCRIPTION:
Two variations of gastric bypass are compared:

Method 1 (test method):A 200 cm BP-limb (distance Treitz to EA) + 150 cm common channel (EA to ileocecal valve) + Roux-Y-limb variable Method 2 (standard method): A 60 cm BP limb + 150 cm Roux-Y-limb + common channel variable.

Patients are evaluated according to the principles of the Scandinavian Obesity surgery registry (SOReg) with the addition of two additional questionnaires.

FU time is set at 5 years.

ELIGIBILITY:
Inclusion Criteria:

* BMI 50-65
* Age 18-55
* Conservative attempts at weight reduction failed

Exclusion Criteria:

* Inability to speak and understand the Swedish language
* Residence outside the county of Skåne
* Psychotic disease
* Inflammatory bowel disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2011-08-29 (Actual); Primary Completion 2015-11-20 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
body weight reduction | 5 years
  absolute BW reduction, percentage of patients reaching BMI below 30,

SECONDARY OUTCOMES:
gastrointestinal function | 5 years
  SF-36, Op-9, GSRS and TFEQ are used in patient assessed variables

CONTACTS AND LOCATIONS:
Overall Officials: Jan L Hedenbro, Principal Investigator — Lunds Universitets Diabetescentrum
Locations (1):
- Aleris Obesity Skåne, Lund, Sweden

REFERENCES:
- [Derived] Nergard BJ, Leifson BG, Gislason H, Hedenbro JL. Effect of different limb lengths on quality of life, eating patterns and gastrointestinal symptoms after Roux-en-Y gastric bypass in superobese patients: randomized study. BJS Open. 2020 Sep 15;4(6):1109-16. doi: 10.1002/bjs5.50334. Online ahead of print. PMID 32931641
- [Derived] Nergard BJ, Lindqvist A, Gislason HG, Groop L, Ekelund M, Wierup N, Hedenbro JL. Mucosal glucagon-like peptide-1 and glucose-dependent insulinotropic polypeptide cell numbers in the super-obese human foregut after gastric bypass. Surg Obes Relat Dis. 2015 Nov-Dec;11(6):1237-46. doi: 10.1016/j.soard.2015.03.021. Epub 2015 Apr 2. PMID 26143297